CLINICAL TRIAL: NCT00003193
Title: Phase I/II Study of Escalating Doses of Taxol Used Concurrently With Ethyol and Accelerated Hyperfractionated Radiotherapy in the Treatment of Stage III and IV Carcinoma of the Head and Neck
Brief Title: Paclitaxel and Radiation Therapy Plus Chemoprotection With Amifostine in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Philip C. Amrein, M.D., Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066028; MGH-M7-20; ALZA-97-024-ii; NCI-V98-1384
Record Dates: First submitted 1999-11-01; First posted 2003-04-23 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Head and Neck Cancer; Oral Complications
Keywords: oral complications; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Amifostine; Paclitaxel; Radiotherapy

ARMS (1):
- Paclitaxel, amifostine, RT (Experimental): Dose-escalation arm for paclitaxel with amifostine and RT.
  Interventions: Drug: amifostine trihydrate; Drug: paclitaxel; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: paclitaxel
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Chemoprotective drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy.

PURPOSE: Phase I/II trial to study the effectiveness of paclitaxel and radiation therapy plus chemoprotection with amifostine in treating patients with stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of paclitaxel with amifostine and radiotherapy in patients with stage III or IV head and neck cancer.
* Determine the toxic effects and complications of this regimen in terms of mucositis reduction in these patients.
* Determine the complete response rate and progression-free survival of patients treated with this regimen.
* Determine whether amifostine modulates the plasma pharmacokinetics of paclitaxel in these patients.

OUTLINE: This is a dose-escalation study of paclitaxel with and without amifostine.

Patients receive paclitaxel IV on days 1, 8, 15, 29, 36, and 43 for a total of 3-6 doses. Patients also undergo radiotherapy twice daily for 6 weeks, except for days when paclitaxel is given.

Cohorts of 2-5 patients receive escalating doses of paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2-3 patients experience dose-limiting toxicity. An additional 10 patients are treated at the MTD.

After determination of the MTD for paclitaxel, subsequent patients also receive amifostine IV over 15 minutes on days 1, 8, 29, and 36 and radiotherapy on days 2-5 and 30-33. Determination of the MTD for this drug combination is carried out as with paclitaxel alone.

At 4 to 8 weeks after the last treatment of radiotherapy, patients undergo CT scanning to determine response. Patients with residual masses undergo neck dissection. Patients with complete or partial response at the primary site are followed without surgery.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A maximum of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III or IV squamous cell head and neck cancer

  * T3-4, N0-3, M0

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance Status:

* ECOG 0-2

Life Expectancy:

* Not specified

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 3.0 mg/dL
* SGOT no greater than 3 times upper limit of normal

Renal:

* Creatinine no greater than 3.0 mg/dL

Other:

* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent beta-adrenergic blocking agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 1998-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months
  Safety is evaluated in this dose-escalation study

SECONDARY OUTCOMES:
Response rate | 6 months
  Response in terms of CR, PR, stable disease, or progression was determined

OTHER OUTCOMES:
Survival | 5 years
  Percentage of patients alive at 5 years as well as the median overal survival were determined.

CONTACTS AND LOCATIONS:
Overall Officials: Philip C. Amrein, MD, Study Chair — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Amrein PC, Clark JR, Supko JG, Fabian RL, Wang CC, Colevas AD, Posner MR, Deschler DG, Rocco JW, Finkelstein DM, McIntyre JF. Phase I trial and pharmacokinetics of escalating doses of paclitaxel and concurrent hyperfractionated radiotherapy with or without amifostine in patients with advanced head and neck carcinoma. Cancer. 2005 Oct 1;104(7):1418-27. doi: 10.1002/cncr.21312. PMID 16116597